CLINICAL TRIAL: NCT06028867
Title: Validation of the Clinical and Antimicrobial Effectiveness of a Clorexidine and Sodium DNA Based Mouthwash in Patients With Stage III and IV Periodontitis: a Randomized-controlled Clinical Trial
Brief Title: Validation of the Clinical and Antimicrobial Effectiveness of a Clorexidine and Sodium DNA Based Mouthwash in Patients With Stage III and IV Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121-29
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: The study was designed as a double-blind randomized controlled trial (RCT) with three parallel groups of individuals.
Who Masked: Participant, Care Provider
Masking Description: Sealed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chlorhexidine 0,12% + Sodium DNA mouthwash (Experimental): Patients are treated with a mouthwash containing Chlorhexidine 0,12% + Sodium DNA
  Interventions: Procedure: Non-surgical periodontal treatment
- Chlorhexidine 0,20% mouthwash (Active Comparator): Patients are treated with a mouthwash containing Chlorhexidine 0,20%
  Interventions: Procedure: Non-surgical periodontal treatment
- Placebo mouthwash (Placebo Comparator): Patients are treated with a placebo mouthwash
  Interventions: Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Subgingival biofilm ultrasonic debridement

SUMMARY:
Sodium DNA has several properties that may be beneficial in the management of bacterial biofilm in periodontitis. The aim of this RCT study is to clinically evaluate the antimicrobial and oral biofilm control properties of two mouthwashes containing Chlorhexidine 0.12% + Sodium DNA and Chlorhexidine 0.20% at two weeks, compared with a placebo, on patients with stage III or IV periodontitis.

DETAILED DESCRIPTION:
Sodium DNA has several properties that may be beneficial in the management of bacterial biofilm in periodontitis. The aim of this RCTstudy is to clinically evaluate the antimicrobial and oral biofilm control properties of two mouthwashes containing Chlorhexidine 0.12% + Sodium DNA and Chlorhexidine 0.20% at two weeks, compared with a placebo, on patients with stage III or IV periodontitis. The study was designed as a double-blind randomized controlled trial (RCT) with three parallel groups of individuals.

ELIGIBILITY:
Inclusion Criteria:

• Clinically diagnosed with stage III or IV periodontitis according to the EFP/AAP 2017 criteria.

Exclusion Criteria:

* Periodontal treatment, antibiotics, NSAIDs, immunosuppressants during the last 6 months.
* Pregnancy.
* Systemic diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Subgingival biofilm | 2 weeks
  Subgingival biofilm collected with sterile paper strips and analyzed by polimerase chain reaction

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: No